CLINICAL TRIAL: NCT03322163
Title: Preconception Maternal Iodine Status and Offspring Cognitive Function: Longitudinal Analyses in the Southampton Women's Survey
Brief Title: Preconception Maternal Iodine Status and Offspring Cognitive Function:
Status: Completed | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: Iodine*CogFn
Record Dates: First submitted 2017-10-11; First posted 2017-10-26 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Cognitive Function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine samples from women collected before they became pregnant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Exposure is maternal iodine — The exposure is preconception maternal iodine status There is no intervention in this observational study

SUMMARY:
Little is known about maternal iodine nutrition before conception and its relation with the child's cognitive function. Using samples and data from the Southampton Women's Survey, iodine measurements from urine collected before the mothers became pregnant will be related to cognitive function measures in the children at age 6-7 years.

DETAILED DESCRIPTION:
Adverse effects of severe maternal iodine deficiency in pregnancy on fetal brain development are well-established, but the effects of mild or moderate deficiency are not well understood. To date, most studies have examined iodine status in pregnancy; less is known about maternal iodine nutrition before conception, and this study aims to address that gap in information

The Southampton Women's Survey (SWS) is a prospective study of mothers and children, established in 1998. A general population sample of 12,583 non-pregnant women, aged 20-34 years resident in Southampton was recruited (1998-2002). All women were visited at home by a research nurse and characterised in detail, including assessments of diet, lifestyle and body composition. Between 1998 and 2007, 3158 of the SWS women became pregnant, and went on to deliver a live singleton infant. These women were followed up in through pregnancy and their children have been assessed in a number of follow-up studies in infancy and childhood. These have included repeated assessments of diet, anthropometry and body composition, as well as detailed functional measurements at specific ages, and are ongoing.

At the 6-7 year assessment, the children's cognitive function was measured and this is the primary outcome.

Spot urine samples were collected from the SWS women at clinic visits following their initial interviews (median 33 (IQR 15-87) days), in the period before conception. The time of day was recorded for each urine collection. Urine samples were split divided into aliquots on the day of collection. They were frozen and stored at -80⁰oC from the date of collection until being thawed and assayed for iodine and creatinine contents in 2016 by the Trace Element Unit, Southampton General NHS Trust Hospital, Southampton, UK.

ELIGIBILITY:
Inclusion Criteria:

* Offspring of women recruited to the Southampton Women's Survey
* Aged 6-7 years at time of measurement

Exclusion Criteria:

* Mother had not provided urine sample before conception of the child

Ages: 6 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The children are part of a cohort study that recruited their mothers before they were conceived. Women registered with a general practitioner in the Southampton area were recruited at ages 20-34 years when they were not pregnant. Those who subsequently became pregnant were followed through the pregnancy and then the children are being followed-up. This study focuses on iodine measures from the preconception recruitment and the follow-up in their homes of the children aged 6-7 years.
Sampling Method: Non-Probability Sample
Enrollment: 12583 (Actual)
Dates: Start 1998-04-06 (Actual); Primary Completion 2014-12-29 (Actual); Study Completion 2014-12-29 (Actual)

PRIMARY OUTCOMES:
Cognitive function | Age 6-7 years
  Cognitive function assessed using the 2-subtest form of the Wechsler Abbreviated Scale of Intelligence and specific components of executive function (Delayed Matching to Subject (DMS), Spatial Span (SSP) and Intra-Extra Dimensional Set Shift (IED)) from the Cambridge Neuropsychological Test Automated Battery (CANTAB®, Cambridge Cognition, Cambridge, UK)

CONTACTS AND LOCATIONS:
Overall Officials: Hazel M Inskip, PhD, Study Director — Deputy Director
Locations (1):
- MRC Lifecourse Epidemiology Unit, University of Southampton, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data from the whole Southampton Women's Survey are shared with other researchers in a collaborative model. Contact can be made via the website: www.mrc.soton.ac.uk
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available once confidentiality arrangements are in place. There is no time restriction.
Access Criteria: See website below.
URL: http://www.mrc.soton.ac.uk

REFERENCES:
- [Background] Inskip HM, Godfrey KM, Robinson SM, Law CM, Barker DJ, Cooper C; SWS Study Group. Cohort profile: The Southampton Women's Survey. Int J Epidemiol. 2006 Feb;35(1):42-8. doi: 10.1093/ije/dyi202. Epub 2005 Sep 29. No abstract available. PMID 16195252